CLINICAL TRIAL: NCT02671435
Title: A Phase 1/2 Study of Durvalumab and Monalizumab in Adult Subjects With Select Advanced Solid Tumors
Brief Title: A Study of Durvalumab (MEDI4736) and Monalizumab in Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419NC00001; D419NC00001 (Other Grant/Funding Number: Medimmune LLC); 2016-000662-38 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Results first posted 2023-03-09 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors
Keywords: Colorectal, colon, CRC, solid tumors, check point inhibitors, immunotherapy, metastatic
MeSH Terms: conditions — Neoplasm Metastasis | interventions — monalizumab; durvalumab; Cetuximab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (15):
- Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W (Experimental): Participants will receive intravenous (IV) infusions of durvalumab 1500 mg every 4 weeks (Q4W) in combination with monalizumab 22.5 mg every 2 weeks (Q2W) up to 3 years until unacceptable toxicity, documentation of confirmed disease progression (PD), or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W (Experimental): Participants will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 75 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W (Experimental): Participants will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 225 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Experimental): Participants will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W (Experimental): Participants will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q4W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) (Experimental): Participants with microsatellite-stable colorectal cancer (MSS-CRC) will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (ovarian) (Experimental): Participants with ovarian cancer will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) (Experimental): Participants with endometrial MSS will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) (Experimental): Participants with non-small cell lung cancer (NSCLC) will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab
- Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W (Experimental): Participants with first-line (1L) MSS-CRC will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W plus mFOLFOX (oxaliplatin 85 mg/m^2 IV infusion, folinic acid 400 mg/m^2 infusion, fluorouracil 400 mg/m^2 IV bolus, followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours on Day 1) Q2W plus IV infusion of bevacizumab 5 mg/kg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab; Drug: mFOLFOX6; Drug: Bevacizumab
- Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W (Experimental): Participants with 1L MSS-CRC will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W, plus mFOLFOX6 (oxaliplatin 85 mg/m^2, folinic acid 400 mg/m^2, fluorouracil 400 mg/m^2 IV bolus, followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours on Day 1) Q2W plus IV infusion of cetuximab (loading dose of 400 mg/m^2 on Day 1, followed by maintenance dose of 250 mg/m^2 IV infusion every week starting on Day 8, then changed to 500 mg/m^2 IV infusion Q2W) up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab; Drug: Cetuximab; Drug: mFOLFOX6
- Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W (Experimental): Participants with recurrent or metastatic third-line (3L) RAS mutant MSS-CRC will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab; Drug: Cetuximab
- Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W (Experimental): Participants with recurrent or metastatic 3L RAS mutant MSS-CRC will receive IV infusion of monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Cetuximab
- Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W (Experimental): Participants with recurrent or metastatic 3L RAS/BRAF wild type MSS-CRC will receive IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Durvalumab; Drug: Cetuximab
- Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W (Experimental): Participants with recurrent or metastatic 3L RAS/BRAF wild type MSS-CRC will receive IV infusion of monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
  Interventions: Drug: Monalizumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Monalizumab — Participants will receive IV infusion of monalizumab as stated in arm description.
Drug: Durvalumab — Participants will receive IV infusion of durvalumab as stated in arm description.
  Arms: Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W; Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W; Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W; Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W; Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W; Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS); Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC); Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC); Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (ovarian); Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W; Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W; Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W; Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W
Drug: Cetuximab — Participants will receive IV infusion of cetuximab as stated in arm description.
  Arms: Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W; Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W; Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W; Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W; Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W
Drug: mFOLFOX6 — Participants will receive IV infusion of mFOLFOX as stated in arm description.
  Arms: Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W; Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W
Drug: Bevacizumab — Participants will receive IV infusion of bevacizumab as stated in arm description.
  Arms: Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W

SUMMARY:
This is a multicenter, open-label, dose-escalation, dose-exploration and dose-expansion study to evaluate the safety, tolerability, antitumor activity, pharmacokinetic (PK), pharmacodynamics, and immunogenicity of durvalumab (MEDI4736) in combination with monalizumab (IPH2201) in adult participants with selected advanced solid tumors and the combination of durvalumab and monalizumab (IPH2201) standard of care systemic therapy with or without biological agent and monalizumab (IPH2201) with biological agent administered to participants with recurrent or metastatic colorectal cancer (CRC).

DETAILED DESCRIPTION:
The study consists of 3 parts: dose escalation (Part 1), dose expansion (Part 2), and dose exploration (Part 3). Part 1 will evaluate dose escalation of durvalumab in combination with monalizumab in adult participants with select advanced solid tumor malignancies. Part 2 will evaluate further the identified dose of durvalumab in combination with monalizumab from Part 1 in adult participants with select advanced solid tumor malignancies. Part 3 will evaluate dose exploration of durvalumab in combination with monalizumab and standard of care systemic therapy with or without biological agent, and monalizumab in combination with biological agent in adult participants with CRC.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologic documentation of advanced recurrent or metastatic cancer.
2. Participants must be at the recurrent/metastatic setting, with selected advanced solid tumors.
3. Participants must have at least one lesion that is measurable by RECIST v1.1
4. Part 3, Dose exploration, CRC participants can be treatment naïve but should not have received more than two line of systemic therapy in the recurrent/metastatic setting.

Exclusion Criteria

1. Prior treatment with immunotherapy agents. Prior treatment with antitumor vaccines may be permitted upon discussion with the medical monitor.
2. Prior participation in clinical studies that include durvalumab alone or in combination, where the study has registrational intent and the analyses for the primary endpoint have not yet been completed
3. Receipt of any conventional or investigational anticancer therapy within 4 weeks prior to the first dose of study treatment
4. Any concurrent chemotherapy, immunotherapy, biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions is acceptable.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 383 (Actual)
Dates: Start 2016-02-22 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2025-09-01 (Estimated)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (22):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Duarte, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, Sacramento, California
  - Research Site, Santa Monica, California
  - Research Site, Aurora, Colorado
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, New Brunswick, New Jersey
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Providence, Rhode Island
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
- Australia (3):
  - Research Site, Blacktown
  - Research Site, Clayton
  - Research Site, Waratah
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Leuven
- Canada (2):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
- France (2):
  - Research Site, Marseille
  - Research Site, Nantes
- Research Site, Debrecen, Hungary
- Research Site, Milan, Italy
- Research Site, Grafton, New Zealand
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Seville
- United Kingdom (2):
  - Research Site, London
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Patel SP, Alonso-Gordoa T, Banerjee S, Wang D, Naidoo J, Standifer NE, Palmer DC, Cheng LY, Kourtesis P, Ascierto ML, Das M, Diamond JR, Hellmann MD, Carneiro BA. Phase 1/2 study of monalizumab plus durvalumab in patients with advanced solid tumors. J Immunother Cancer. 2024 Feb 2;12(2):e007340. doi: 10.1136/jitc-2023-007340. PMID 38309722
- [Derived] Hwang M, Fan C, Yue MS, Zhou D, Paturel C, Andre P, Cheng LY, Mitchell P, Kourtesis P, Ruscica D, Das M, Morsli N, Ren S, Gibbs M, Phipps A, Song X. Population Pharmacokinetics of Monalizumab in Patients With Advanced Solid Tumors. J Clin Pharmacol. 2023 Jul;63(7):817-829. doi: 10.1002/jcph.2220. Epub 2023 Apr 10. PMID 36852723
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419NC00001&attachmentIdentifier=0025c0b0-10b2-4c30-a0be-d095e7e9d3a6&fileName=D419NC00001_Amd_6_Protocol_(1)-Redacted.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419NC00001&attachmentIdentifier=d3f8249c-94ba-4dbd-b4a1-626d65c0860d&fileName=d419nc00001-sap-ed-2-Redacted.pdf&versionIdentifier=
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419NC00001&attachmentIdentifier=355cf93c-e8f1-452b-8fff-50f057aa7eee&fileName=D419NC00001_CSR_Synopsis_(21Sep22)-Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W: Participants received intravenous (IV) infusions of durvalumab 1500 mg every 4 weeks (Q4W) in combination with monalizumab 22.5 mg every 2 weeks (Q2W) up to 3 years until unacceptable toxicity, documentation of confirmed disease progression (PD), or documentation of subject withdrawal for another reason.
- Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W: Participants received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 75 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W: Participants received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 225 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W: Participants received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W: Participants received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q4W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC): Participants with microsatellite-stable colorectal cancer (MSS-CRC) received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian): Participants with ovarian cancer received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS): Participants with endometrial MSS received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC): Participants with non-small cell lung cancer (NSCLC) received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W: Participants with first-line (1L) MSS-CRC received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W plus mFOLFOX (oxaliplatin 85 mg/m^2 IV infusion, folinic acid 400 mg/m^2 infusion, fluorouracil 400 mg/m^2 IV bolus, followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours on Day 1) Q2W plus IV infusion of bevacizumab 5 mg/kg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W: Participants with 1L MSS-CRC received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W, plus mFOLFOX6 (oxaliplatin 85 mg/m^2, folinic acid 400 mg/m^2, fluorouracil 400 mg/m^2 IV bolus, followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours on Day 1) Q2W plus IV infusion of cetuximab (loading dose of 400 mg/m^2 on Day 1, followed by maintenance dose of 250 mg/m^2 IV infusion every week starting on Day 8, then changed to 500 mg/m^2 IV infusion Q2W) up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W: Participants with recurrent or metastatic third-line (3L) RAS mutant MSS-CRC received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W: Participants with recurrent or metastatic 3L RAS mutant MSS-CRC received IV infusion of monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W: Participants with recurrent or metastatic 3L RAS/BRAF wild type MSS-CRC received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W: Participants with recurrent or metastatic 3L RAS/BRAF wild type MSS-CRC received IV infusion of monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
Period: Overall Study
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Started | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 40 | 41 | 44 | 37
Treated | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 37
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 40 | 41 | 44 | 37
Not completed — Death | 1 | 3 | 0 | 16 | 14 | 29 | 34 | 28 | 19 | 10 | 8 | 29 | 29 | 29 | 27
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 2 | 0 | 2 | 0 | 3 | 3 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 2 | 2 | 7 | 2 | 7 | 1 | 1 | 2 | 4 | 4 | 4 | 2
Not completed — Un-specified | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 3 | 0 | 5 | 8 | 4 | 5 | 9 | 8

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included participants who were randomized and were analyzed according to the treatment group they were randomized to.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Total
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 40 | 41 | 44 | 37 | 383
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (21.7) | 55.7 (18.0) | 59 (15.1) | 56.4 (13.5) | 60 (13.5) | 53.6 (12.9) | 61.5 (9.1) | 63.7 (8.5) | 63.2 (7.9) | 60.8 (9.9) | 55.4 (9.4) | 55.8 (10.7) | 52.3 (10.6) | 55.9 (11.3) | 58.8 (9.6) | 57.8 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 2 | 17 | 6 | 15 | 40 | 40 | 6 | 8 | 8 | 17 | 16 | 17 | 18 | 216
  Male | 0 | 0 | 1 | 1 | 12 | 25 | 0 | 0 | 14 | 10 | 10 | 23 | 25 | 27 | 19 | 167
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 3 | 0 | 6 | 5 | 3 | 2 | 1 | 1 | 3 | 6 | 4 | 0 | 36
  Not Hispanic or Latino | 2 | 2 | 3 | 15 | 17 | 34 | 35 | 37 | 16 | 17 | 17 | 37 | 35 | 40 | 37 | 344
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 2 | 3 | 1 | 2 | 0 | 1 | 4 | 9 | 8 | 14 | 13 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3
  Black or African American | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 4 | 1 | 2 | 0 | 2 | 1 | 1 | 1 | 17
  White | 3 | 3 | 3 | 15 | 15 | 36 | 35 | 30 | 16 | 13 | 13 | 29 | 30 | 25 | 22 | 288
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 2 | 2 | 1 | 0 | 2 | 2 | 1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug. Any TEAEs data is inclusive of both serious and other adverse events (non-serious).
Time Frame: Day 1 through 246.9 weeks (maximum observed duration)
Population: As-treated population included participants who received any study drugs and were analyzed according to the treatment they actually received.
Measure: Count of Participants; unit: Participants
Groups:
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC): Participants with MSS-CRC received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC): Participants with NSCLC received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 37
Participants
  Any TEAEs | 3 | 3 | 3 | 18 | 17 | 39 | 40 | 39 | 20 | 18 | 18 | 39 | 41 | 44 | 36
  Any TESAEs | 1 | 0 | 1 | 8 | 4 | 11 | 16 | 17 | 7 | 10 | 11 | 10 | 5 | 9 | 11

2. Primary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Change from baseline in SBP and DBP (minimum post baseline change [PBC] and maximum PBC) are reported.
Time Frame: Day 1 (baseline) through 246.9 weeks (maximum observed duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 37
mmHg
  SBP min PBC | -19.00 (21.63) | -26.00 (10.82) | -14.67 (11.55) | -22.94 (12.73) | -23.06 (20.48) | -21.45 (12.89) | -22.55 (13.35) | -21.23 (12.29) | -26.40 (12.75) | -29.28 (19.19) | -24.61 (10.92) | -23.31 (12.88) | -20.80 (11.87) | -25.57 (13.99) | -25.05 (16.86)
  SBP max PBC | 27.33 (5.69) | 19.00 (5.57) | 28.67 (20.82) | 29.22 (15.78) | 22.00 (19.16) | 21.10 (12.04) | 22.15 (17.39) | 23.55 (14.13) | 22.95 (11.69) | 27.17 (21.63) | 23.61 (11.27) | 20.74 (15.31) | 17.20 (10.51) | 23.00 (13.18) | 22.59 (15.69)
  DBP min PBC | -15.67 (18.01) | -22.00 (10.00) | -10.67 (9.07) | -17.89 (9.58) | -18.61 (11.05) | -16.60 (10.40) | -17.60 (9.81) | -13.05 (7.21) | -19.15 (10.28) | -18.11 (8.98) | -20.50 (9.79) | -16.13 (9.33) | -16.39 (9.94) | -18.09 (9.69) | -17.68 (12.15)
  DBP max PBC | 23.67 (11.93) | 11.67 (4.93) | 18.00 (9.64) | 14.06 (12.75) | 12.39 (9.30) | 15.58 (9.69) | 12.63 (11.11) | 19.83 (10.15) | 16.65 (9.46) | 18.11 (9.33) | 14.22 (12.18) | 13.54 (10.01) | 13.10 (8.98) | 16.05 (10.06) | 14.43 (9.01)

3. Primary Outcome: Change From Baseline in Respiratory Rate (RR)
Description: Change from baseline in RR (minimum PBC and maximum PBC) are reported.
Time Frame: Day 1 (baseline) through 246.9 weeks (maximum observed duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 37
breaths/min
  RR min PBC | -2.00 (2.00) | -3.00 (1.00) | -1.33 (2.31) | -1.78 (1.31) | -1.50 (1.86) | -1.93 (1.86) | -1.53 (1.52) | -1.83 (1.62) | -1.55 (3.12) | -2.00 (1.94) | -1.67 (1.78) | -2.15 (2.23) | -1.59 (1.52) | -2.00 (1.33) | -1.92 (1.89)
  RR max PBC | 2.00 (3.46) | 2.33 (0.58) | 2.67 (1.15) | 1.72 (1.49) | 1.83 (1.42) | 2.40 (2.37) | 2.53 (2.24) | 2.40 (2.62) | 4.05 (3.09) | 2.50 (2.09) | 3.39 (3.62) | 1.85 (1.73) | 2.00 (1.55) | 2.59 (1.83) | 3.14 (4.60)

4. Primary Outcome: Change From Baseline in Pulse Rate (PR)
Description: Change from baseline in PR (minimum PBC and maximum PBC) are reported.
Time Frame: Day 1 (baseline) through 246.9 weeks (maximum observed duration)
Population: As-treated population included participants who received any study drugs and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 38 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 37
beats/min
  PR min PBC | -5.33 (2.52) | -14.33 (6.51) | -7.00 (1.73) | -15.67 (11.83) | -15.39 (9.20) | -14.70 (9.39) | -12.24 (10.10) | -11.38 (10.98) | -13.95 (9.12) | -15.67 (8.84) | -18.11 (11.98) | -15.74 (11.20) | -13.15 (11.89) | -13.91 (7.04) | -11.68 (9.02)
  PR max PBC | 38.33 (10.02) | 16.67 (6.11) | 21.67 (8.08) | 19.33 (15.05) | 17.78 (11.12) | 20.28 (10.03) | 20.68 (13.42) | 22.60 (12.17) | 25.80 (11.27) | 21.28 (13.48) | 21.06 (12.24) | 23.54 (12.83) | 23.88 (11.31) | 25.18 (13.71) | 27.38 (13.92)

5. Primary Outcome: Change From Baseline in Body Temperature (BT)
Description: Change from baseline in BT (minimum PBC and maximum PBC) are reported.
Time Frame: Day 1 (baseline) through 246.9 weeks (maximum observed duration)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 37
degree Celsius
  BT min PBC | -0.30 (0.30) | -0.37 (0.38) | -0.67 (0.55) | -0.66 (0.56) | -0.48 (0.28) | -0.62 (0.39) | -0.63 (0.42) | -0.47 (0.32) | -0.51 (0.26) | -0.84 (0.46) | -0.79 (0.48) | -0.51 (0.39) | -0.52 (0.33) | -0.65 (0.45) | -0.66 (0.58)
  BT max PBC | 0.63 (0.32) | 0.93 (0.92) | 0.50 (0.26) | 0.78 (0.72) | 0.60 (0.73) | 0.65 (0.43) | 0.64 (0.46) | 0.77 (0.47) | 0.72 (0.46) | 0.89 (0.51) | 0.56 (0.43) | 0.75 (0.57) | 0.70 (0.53) | 0.91 (0.64) | 0.81 (0.66)

6. Primary Outcome: Change From Baseline in Oxygen Saturation (OS)
Description: Change from baseline in OS (minimum PBC and maximum PBC) are reported.
Time Frame: Day 1 (baseline) through 246.9 weeks (maximum observed duration)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of oxygen saturation
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 0 | 1 | 2 | 1 | 0 | 2 | 1 | 6
Percentage of oxygen saturation
  OS min PBC | -1.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. |  |  | -3.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. | -3.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. | -0.67 (1.53) | -21.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. |  | 0 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. | 0.50 (2.12) | -4.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. |  | 0.50 (0.71) | -1.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. | -0.33 (2.80)
  OS max PBC | -1.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. |  |  | -3.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. | -3.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. | -0.67 (1.53) | -21.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. |  | 0 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. | 0.50 (2.12) | -4.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. |  | 0.50 (0.71) | -1.00 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm group. | -0.33 (2.80)

7. Primary Outcome: Number of Participants With Notable Change in QTcF and QTcB From Baseline
Description: Participants who had notable QTcF and QTcB interval change from baseline are reported.
Time Frame: Day 1 (baseline) through 246.9 weeks (maximum observed duration)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 16 | 18 | 39 | 38 | 40 | 19 | 18 | 17 | 39 | 40 | 43 | 37
Participants
  QTcF>30 msec | 0 | 0 | 0 | 2 | 1 | 6 | 5 | 2 | 2 | 1 | 2 | 3 | 3 | 5 | 5
  QTcF>60 msec | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1
  QTcB>30 msec | 1 | 0 | 0 | 3 | 2 | 5 | 5 | 4 | 3 | 1 | 6 | 4 | 8 | 9 | 6
  QTcB>60 msec | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1

8. Primary Outcome: Number of Participants With at Least 2-Grade Shift From Baseline in Laboratory Parameters
Description: Number of participants with at least 2-Grade shift from baseline in laboratory parameters are reported.
Time Frame: Day 1 (baseline) through 246.9 weeks (maximum observed duration)
Population: As-treated population included participants who received any study drugs and were analyzed according to the treatment they actually received. Here, number analyzed (n) denotes number of participants analyzed for the specified laboratory parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 37
Participants
  Anaemia: number analyzed (Participants) | 3 | 3 | 3 | 17 | 18 | 40 | 38 | 38 | 20 | 17 | 18 | 39 | 41 | 44 | 37
  Anaemia | 0 | 0 | 1 | 2 | 1 | 2 | 1 | 2 | 0 | 1 | 2 | 2 | 2 | 0 | 2
  White blood cell decreased: number analyzed (Participants) | 3 | 3 | 3 | 17 | 18 | 40 | 38 | 38 | 20 | 17 | 18 | 39 | 41 | 44 | 37
  White blood cell decreased | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 7 | 6 | 0 | 2 | 4 | 1
  Lymphocyte count decreased: number analyzed (Participants) | 3 | 3 | 3 | 17 | 18 | 40 | 38 | 38 | 20 | 17 | 18 | 39 | 41 | 44 | 37
  Lymphocyte count decreased | 0 | 1 | 1 | 4 | 4 | 5 | 7 | 8 | 5 | 5 | 4 | 6 | 3 | 7 | 8
  Lymphocyte count increased: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 17 | 18 | 39 | 41 | 44 | 37
  Lymphocyte count increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Neutrophil count decreased: number analyzed (Participants) | 3 | 3 | 3 | 17 | 18 | 40 | 38 | 38 | 20 | 17 | 18 | 37 | 37 | 36 | 31
  Neutrophil count decreased | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 9 | 11 | 0 | 1 | 1 | 1
  Platelet count decreased: number analyzed (Participants) | 3 | 3 | 3 | 17 | 18 | 40 | 38 | 38 | 20 | 17 | 18 | 39 | 41 | 43 | 37
  Platelet count decreased | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 0 | 0 | 3
  Hypoalbuminemia: number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 36
  Hypoalbuminemia | 1 | 0 | 0 | 6 | 3 | 6 | 6 | 6 | 2 | 2 | 2 | 9 | 2 | 6 | 5
  Creatinine increased: number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 0 | 0 | 0 | 0
  Creatinine increased | 1 | 1 | 1 | 1 | 4 | 4 | 4 | 8 | 2 | 4 | 2 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase increased: number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Gamma Glutamyl Transferase increased | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia: number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 0 | 0 | 0 | 0
  Hyponatremia | 1 | 0 | 1 | 2 | 3 | 3 | 5 | 5 | 1 | 4 | 2 | 0 | 0 | 0 | 0
  Hyperglycemia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 40 | 40 | 40 | 20 | 18 | 18 | 0 | 0 | 0 | 0
  Hyperglycemia | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 3 | 5 | 1 | 5 | 0 | 0 | 0 | 0
  Serum amylase increased: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0 | 0 | 0
  Serum amylase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 6 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0 | 0 | 0
  Aspartate aminotransferase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
  Blood bilirubin increased: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 39 | 40 | 43 | 37
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 7 | 7 | 3 | 6
  Lipase increased: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 39 | 40 | 44 | 36
  Lipase increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 10 | 5 | 6 | 7 | 5
  Hypertriglyceridemia: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 18 | 18 | 0 | 0 | 0 | 0
  Hypertriglyceridemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 0 | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLT: Any study drug related Grade (G) 3 or higher toxicity that occurred during DLT evaluation period including: any G>=3 noninfectious colitis/pneumonitis, liver transaminase elevation (TE) >=5 but =<8 upper limit of normal (ULN), any G4 immune-mediated AE (imAE)/immune-related AE (irAE), any G>=3 clinically significant non-hematologic toxicity, TE >8 ULN or total bilirubin (TBL) >5 ULN, increase in AST or ALT >=3 ULN along with TBL >=2 ULN, thrombocytopenia (G3/4 associated with G3/higher hemorrhage, G3 that did not improve by at least 1 grade within 7 days, and G4), G4 febrile neutropenia (FN), G3 FN of >=5 days and G3 FN regardless of duration, G4 neutropenia of >7 days, G3/4 neutropenia not associated with fever/systemic infection, and anemia (G3 and G4).
Time Frame: From Day 1 to 28 days after the first dose of study drugs
Population: The DLT-Evaluable population included all participants enrolled in the dose-escalation part who received at least 1 dose of study drugs and completed the safety follow-up through the DLT-evaluation period or experienced any DLT during the DLT-evaluation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W
Number analyzed (Participants) | 3 | 3 | 3 | 17 | 18
Participants | 0 | 0 | 0 | 0 | 0

10. Primary Outcome: Percentage of Participants With Objective Response (OR) in Exploration Cohorts C1A and C1B
Description: The OR is defined as best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumours Version 1.1 (RECIST V 1.1) guidelines. The CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in between.
Time Frame: Baseline (Days -28 to -1) through 54.8 months (maximum observed duration)
Population: The ITT population included participants who were randomized and were analyzed according to the treatment group they were randomized to.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 40 | 41
Percentage of Participants | 0 [0.0 to 10.3] | 0 [0.0 to 9.0]

11. Secondary Outcome: Percentage of Participants With OR
Description: The OR is defined as best overall response of CR or confirmed PR according to RECIST V 1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in between.
Time Frame: Baseline (Days -28 to -1) through 54.8 months (maximum observed duration)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18
Percentage of Participants | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 84.2] | 0 [0.0 to 19.5] | 0 [0.0 to 19.5] | 7.5 [1.6 to 20.4] | 5.0 [0.7 to 18.2] | 0 [0.0 to 9.5] | 10.0 [1.2 to 31.7] | 44.4 [23.0 to 72.2] | 72.2 [46.5 to 90.3]

12. Secondary Outcome: Percentage of Participants With OR in Exploration Cohorts C2A and C2B
Description: The OR is defined as best overall response of confirmed CR or confirmed PR according to RECIST V 1.1 guidelines. The CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in between.
Time Frame: Baseline (-28 to -1 day) through 54.8 months (maximum observed duration)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 44 | 37
Percentage of Participants | 11.4 [4.0 to 25.6] | 5.4 [0.7 to 18.7]

13. Secondary Outcome: Percentage of Participants With Disease Control (DC)
Description: The DC is defined as best overall response of confirmed CR, confirmed PR, or stable disease (SD) based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in between. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. Participants with SD were included in the DC if they maintained SD for >= 8 weeks from start of treatment. The DCR16 and DCR24 are reported (participants with SD >= 16 weeks and >=24 weeks).
Time Frame: Baseline (-28 to -1 day) through 54.8 months (maximum observed duration)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18
Percentage of Participants
  DCR16 | 0 [0.0 to 70.8] | 33.3 [0.8 to 90.6] | 0 [0.0 to 70.8] | 22.2 [6.4 to 47.6] | 27.8 [9.7 to 53.5] | 30 [16.6 to 46.5] | 30 [16.6 to 46.5] | 25 [12.7 to 41.2] | 40 [19.1 to 63.9] | 77.8 [52.4 to 93.6] | 88.9 [65.3 to 98.6]
  DCR24 | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 18.5] | 11.1 [1.4 to 34.7] | 17.5 [7.3 to 32.8] | 15 [5.7 to 29.8] | 12.5 [4.2 to 26.8] | 25 [8.7 to 49.1] | 66.7 [41.0 to 86.7] | 77.8 [52.4 to 93.6]

14. Secondary Outcome: Percentage of Participants With DC in Exploration Cohorts (C1A, C1B, C2A, and C2B)
Description: The DC is defined as best overall response of confirmed CR, confirmed PR, or SD based on RECIST v1.1. The CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in between. The SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression. Participants with SD were included in the DC if they maintained SD for >= 8 weeks from start of treatment. The DCR16 and DCR24 are reported (participants with SD >= 16 weeks and >=24 weeks).
Time Frame: Baseline (-28 to -1 day) through 54.8 months (maximum observed duration)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 40 | 41 | 44 | 37
Percentage of Participants
  DCR16 | 17.5 [7.3 to 32.8] | 34.1 [20.1 to 50.6] | 59.1 [43.2 to 73.7] | 56.8 [39.5 to 72.9]
  DCR24 | 10.0 [2.8 to 23.7] | 7.3 [1.5 to 19.9] | 52.3 [36.7 to 67.5] | 45.9 [29.5 to 63.1]

15. Secondary Outcome: Duration of Response (DoR)
Description: The DoR is defined as the duration from the first documentation of OR (confirmed CR or confirmed PR) to the first documented disease progression (PD) based on RECIST v1.1 or death due to any cause, whichever occurred first. The CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in between. The PD is defined as at least a 20% increase in the sum of diameters of target lesions or unequivocal progression of existing non-target lesions, taking as reference the smallest sum on study and appearance of one or more new lesions. The DoR was evaluated using Kaplan-Meier method.
Time Frame: Baseline (-28 to -1 day) through 54.8 months (maximum observed duration)
Population: As-treated population included participants who received any study drugs and were analyzed according to the treatment they actually received. Participants who had achieved OR were evaluated for this outcome.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 2 | 8 | 13
Weeks |  |  |  |  |  | 16.1 [15.9 to NA] — Upper limit of 95% confidence interval (CI) could not be derived due to insufficient events being observed. | 68.1 [24.0 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed. |  | 22.9 [10.1 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed. | 66.1 [16.1 to 85.4] | 72.3 [17.4 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed.

16. Secondary Outcome: DoR in Exploration Cohorts (C1A, C1B, C2A, and C2B)
Description: The DoR is defined as the duration from the first documentation of OR (confirmed CR or confirmed PR) to the first documented PD based on RECIST v1.1 or death due to any cause, whichever occurred first. The CR is defined as disappearance of all target and non-target lesions and normalization of tumor marker level lesions. The PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (compared to baseline) and no new nontarget lesion. A confirmed PR is defined as two PRs or an un-confirmed PR and an unconfirmed CR that were separated by at least 28 days with no evidence of progression in between. The PD is defined as at least a 20% increase in the sum of diameters of target lesions or unequivocal progression of existing non-target lesions, taking as reference the smallest sum on study and appearance of one or more new lesions. The DoR was evaluated using Kaplan-Meier method.
Time Frame: Baseline (-28 to -1 day) through 54.8 months (maximum observed duration)
Population: The ITT population included participants who were randomized and were analyzed according to the treatment group they were randomized to. Participants who had achieved OR were evaluated for this outcome.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 0 | 0 | 5 | 2
Weeks |  |  | 32.1 [16.0 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed. | 24.1 [12.1 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed.

17. Secondary Outcome: Progression-Free Survival (PFS)
Description: The PFS is defined as the time from the start of study treatment until the first documentation of PD based on RECIST v1.1 or death due to any cause, whichever occurred first. The PD is defined as at least a 20% increase in the sum of diameters of target lesions or unequivocal progression of existing non-target lesions, taking as reference the smallest sum on study and appearance of one or more new lesions. The PFS was estimated using Kaplan-Meier method.
Time Frame: Baseline (-28 to -1 day) through 54.8 months (maximum observed duration)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18
Months | 1.8 [1.7 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed. | 1.9 [1.8 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed. | 1.9 [NA to NA] — Upper and lower limit of 95% CI could not be derived due to insufficient events being observed. | 2.0 [1.7 to 3.4] | 1.8 [1.7 to 3.5] | 1.9 [1.8 to 3.6] | 1.8 [1.7 to 1.9] | 1.8 [1.7 to 3.3] | 1.9 [1.7 to 3.7] | 10.9 [5.7 to 17.7] | 14.7 [5.8 to 20.9]

18. Secondary Outcome: Progression-Free Survival (PFS) in Exploration Cohorts (C1A, C1B, C2A, and C2B)
Description: as for outcome 17
Time Frame: Baseline (-28 to -1 day) through 54.8 months (maximum observed duration)
Population: as for outcome 10
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 40 | 41 | 44 | 37
Months | 1.8 [1.7 to 1.9] | 2.0 [1.7 to 3.3] | 5.3 [3.2 to 5.5] | 4.4 [2.1 to 5.5]

19. Secondary Outcome: Overall Survival
Description: The overall survival is defined as the time from the start of study treatment until death due to any cause. The overall survival was estimated using Kaplan-Meier method.
Time Frame: Baseline (-28 to -1 day) through 54.8 months (maximum observed duration)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18
Months | 15.1 [NA to NA] — Upper and lower limits of 95% CI could not be derived due to insufficient events being observed. | 20.1 [18.6 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed. | NA [NA to NA] — Median and limits of 95% CI could not be derived due to insufficient events being observed. | 8.1 [4.0 to 16.7] | 13.4 [4.4 to 16.9] | 10.6 [6.0 to 20.1] | 16.7 [10.7 to 21.4] | 11.0 [6.7 to 17.3] | 8.8 [5.8 to 15.6] | 25.6 [13.8 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed. | 29.6 [19.8 to NA] — Upper limit of 95% CI could not be derived due to insufficient events being observed.

20. Secondary Outcome: Overall Survival in Exploration Cohorts (C1A, C1B, C2A, and C2B)
Description: as for outcome 19
Time Frame: Baseline (-28 to -1 day) through 54.8 weeks (maximum observed duration)
Population: The ITT population included participants who were randomized and the participants were analyzed according to the treatment group they were randomized to.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 40 | 41 | 44 | 37
Months | 10.3 [4.3 to 12.7] | 8.9 [6.8 to 11.3] | 14.6 [10.0 to 19.4] | 14.6 [7.2 to 18.7]

21. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Monalizumab
Description: Serum Cmax of monalizumab at pre-dose and end of infusion are reported.
Time Frame: Day 85: Pre-dose and end of infusion (within 10 minutes) after cohort specific infusions
Population: Pharmacokinetic (PK) evaluable population included participants who received at least 1 dose of durvalumab and/or monalizumab and had at least 1 post-treatment sample available. Number of participants analyzed (N) denotes those participants who had adequate PK sample available for analysis. Data for dose-escalation Cohort 4 and dose-expansion Cohorts (MSS-CRC, Ovarian, Endometrial MSS and NSCLC) were combined in a single arm/group to avoid increased variability due to smaller cohort sizes.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Dose-escalation Cohort 4 + Dose-expansion: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W: Participants with solid tumors, microsatellite-stable colorectal cancer (MSS-CRC), ovarian cancer, MSS endometrial cancer or non-small cell lung cancer (NSCLC) received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
- Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W: Participants with recurrent or metastatic 3L RAS mutant MSS-CRC in dose exploration phase received IV infusion of monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15 up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4 + Dose-expansion: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 1 | 2 | 1 | 60 | 6 | 7 | 9 | 10 | 11 | 19 | 19
µg/mL | 7.85 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm. | 43.62 (12.54) | 144.88 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm. | 315.74 (129.08) | 245.18 (142.35) | 304.48 (66.75) | 281.53 (155.57) | 346.85 (91.06) | 388.60 (194.64) | 289.25 (194.59) | 409.93 (175.43)

22. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Monalizumab
Description: Serum Cmin of monalizumab at pre-dose and end of infusion are reported.
Time Frame: Day 85: Pre-dose and end of infusion (within 10 minutes) after cohort specific infusions
Population: Pharmacokinetic evaluable population included participants who received at least 1 dose of durvalumab and/or monalizumab and had at least 1 post-treatment sample available. Number of participants analyzed (N) denotes those participants who had adequate PK sample available for analysis. Data for dose-escalation Cohort 4 and dose-expansion Cohorts (MSS-CRC, Ovarian, Endometrial MSS and NSCLC) were combined in a single arm/group to avoid increased variability due to smaller cohort sizes.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4 + Dose-expansion: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 1 | 2 | 1 | 61 | 6 | 10 | 11 | 11 | 11 | 22 | 22
µg/mL | 7.45 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm. | 18.16 (6.70) | 92.55 (NA) — Standard deviation was not reported as only one participant was evaluable for the specified arm. | 145.04 (76.34) | 67.75 (57.82) | 141.39 (57.01) | 109.18 (45.54) | 129.59 (45.72) | 172.90 (84.55) | 148.05 (70.23) | 185.60 (105.68)

23. Secondary Outcome: Serum Concentration of Durvalumab
Description: Serum concentration of durvalumab is reported.
Time Frame: Pre-dose (PRE) on Day 1 of Weeks 1, 5, 9, 13, and 25 and post-dose (POST) on Day 1 of Weeks 1 and 13
Population: PK evaluable population: Participants who received at least 1 dose of durvalumab and/or monalizumab and had at least 1 post-treatment sample available. Number of participants analyzed (N) denotes those participants who had adequate PK sample for analysis and number analyzed (n) denotes those participants who were analyzed for specified timepoint. Data is combined in a single arm with a respectable sample size as values from different cohorts with small cohort size will increase variability.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Dose-escalation Cohorts(1-5)+Dose-expansion Cohorts+Dose-exploration Cohorts(A1,A2,C1A,C1B,C2A,C2B): Participants in dose-escalation cohorts (1, 2, 3, 4, and 5) received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 22.5, 75, 225 or 750 mg Q2W (Cohorts 1, 2, 3 and 4) or 750 mg Q4W (Cohort 5), dose-expansion cohorts (MSS-CRC, ovarian cancer, MSS endometrial or NSCLC) participants received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W. Participants with recurrent or metastatic 3L RAS mutant (C1A) or RAS/BRAF wild type (C2A) MSS-CRC received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15. Participants with 1L MSS-CRC in Cohorts A1 and A2 received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W, plus mFOLFOX6 (oxaliplatin 85 mg/m^2, folinic acid 400 mg/m^2, fluorouracil 400 mg/m^2 IV bolus, followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours on Day 1) Q2W plus either plus IV infusion of bevacizumab 5 mg/kg Q2W (Cohort A1) or IV infusion of cetuximab (loading dose of 400 mg/m^2 on Day 1, followed by maintenance dose of 250 mg/m^2 IV infusion every week starting on Day 8, then changed to 500 mg/m^2 IV infusion Q2W) (Cohort A2). Participants in all cohorts received treatment up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
Arm/Group | Dose-escalation Cohorts(1-5)+Dose-expansion Cohorts+Dose-exploration Cohorts(A1,A2,C1A,C1B,C2A,C2B)
Number analyzed (Participants) | 287
µg/mL
  Week 1 Day 1 (PRE) | 0.100 (0.63)
  Week 1 Day 1 (POST): number analyzed (Participants) | 285
  Week 1 Day 1 (POST) | 399 (157)
  Week 5 Day 1 (PRE): number analyzed (Participants) | 248
  Week 5 Day 1 (PRE) | 90.8 (95.0)
  Week 9 Day 1 (PRE): number analyzed (Participants) | 193
  Week 9 Day 1 (PRE) | 127 (148)
  Week 13 Day 1 (PRE): number analyzed (Participants) | 140
  Week 13 Day 1 (PRE) | 142 (123)
  Week 13 Day 1 (POST): number analyzed (Participants) | 126
  Week 13 Day 1 (POST) | 497 (277)
  Week 25 Day 1 (PRE): number analyzed (Participants) | 79
  Week 25 Day 1 (PRE) | 149 (109)

24. Secondary Outcome: Serum Concentration of Cetuximab
Description: Serum concentration of cetuximab is reported.
Time Frame: Pre-dose (PRE) on Day 1 of Weeks 1, 5, 9, and 13 and post-dose (POST) on Day 1 of Weeks 1, 5, and 13
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Exploration CohortsA2 (Mona+Durva+mFOLFOX6+Cetu), C1A, C2A (Mona+Durva+Cetu), C1B, C2B (Mona+Cetu): Participants with recurrent or metastatic 3L RAS mutant (C1A) or RAS/BRAF wild type (C2A) MSS-CRC received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15. Participants with recurrent or metastatic 3L RAS mutant (C1B) or RAS/BRAF wild type (C2B) MSS-CRC received IV infusions monalizumab 750 mg Q2W plus IV infusion of cetuximab 500 mg/m^2 on Day 1 then 500 mg/m^2 IV infusion Q2W starting on Day 15. Participants with 1L MSS-CRC in Cohort A2 received IV infusions of durvalumab 1500 mg Q4W in combination with monalizumab 750 mg Q2W, plus mFOLFOX6 (oxaliplatin 85 mg/m^2, folinic acid 400 mg/m^2, fluorouracil 400 mg/m^2 IV bolus, followed by 2400 mg/m^2 continuous IV infusion over 46 to 48 hours on Day 1) Q2W plus IV infusion of cetuximab (loading dose of 400 mg/m^2 on Day 1, followed by maintenance dose of 250 mg/m^2 IV infusion every week starting on Day 8, then changed to 500 mg/m^2 IV infusion Q2W) (Cohort A2). Participants in all cohorts received treatment up to 3 years until unacceptable toxicity, documentation of confirmed PD, or documentation of subject withdrawal for another reason.
Arm/Group | Exploration CohortsA2 (Mona+Durva+mFOLFOX6+Cetu), C1A, C2A (Mona+Durva+Cetu), C1B, C2B (Mona+Cetu)
Number analyzed (Participants) | 70
µg/mL
  Week 1 Day 1 (PRE): number analyzed (Participants) | 54
  Week 1 Day 1 (PRE) | 0.025 (0.00)
  Week 1 Day 1 (POST) | 400 (138)
  Week 5 Day 1 (PRE): number analyzed (Participants) | 48
  Week 5 Day 1 (PRE) | 73.6 (108.0)
  Week 5 Day 1 (POST): number analyzed (Participants) | 6
  Week 5 Day 1 (POST) | 344 (161)
  Week 9 Day 1 (PRE): number analyzed (Participants) | 18
  Week 9 Day 1 (PRE) | 97.7 (137)
  Week 13 Day 1 (PRE): number analyzed (Participants) | 20
  Week 13 Day 1 (PRE) | 61.7 (113)
  Week 13 Day 1 (POST): number analyzed (Participants) | 19
  Week 13 Day 1 (POST) | 387 (101)

25. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibodies (ADA) to Monalizumab
Description: Number of participants with positive ADA to monalizumab are reported. Persistent positive is defined as positive at >= 2 post-baseline assessments (with >=16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive is defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >= 2 post-baseline assessments (with <16 weeks between first and last positive). Treatment-boosted ADA is defined as baseline ADA titer that was boosted to a 4-fold or higher level following drug administration. Treatment-emergent ADA is defined as the sum of treatment-induced ADA (post-baseline positive only) and treatment-boosted ADA.
Time Frame: Day 1 through 54.8 months (Day 1 of Weeks 1, 5, 13, and 25, and 90 days after the last dose of monalizumab)
Population: As-treated population included participants who received any study drugs and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants who had post-baseline ADA results.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 15 | 16 | 36 | 35 | 32 | 18 | 16 | 18 | 30 | 38 | 37 | 34
Participants
  Persistent Positive | 0 | 0 | 0 | 2 | 0 | 10 | 5 | 4 | 2 | 0 | 1 | 5 | 5 | 3 | 5
  Transient Positive | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 1 | 2 | 0
  Treatment-boosted ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-emergent ADA | 0 | 0 | 0 | 3 | 0 | 11 | 7 | 5 | 4 | 0 | 1 | 6 | 6 | 5 | 5

26. Secondary Outcome: Number of Participants With Positive ADA to Durvalumab
Description: Number of participants with positive ADA to monalizumab are reported. Persistent positive is defined as positive at >= 2 post-baseline assessments (with >= 16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive is defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >= 2 post-baseline assessments (with <16 weeks between first and last positive). Treatment-boosted ADA is defined as baseline ADA titer that was boosted to a 4-fold or higher level following drug administration. Treatment-emergent ADA is defined as the sum of treatment-induced ADA (post-baseline positive only) and treatment-boosted ADA.
Time Frame: Day 1 through 54.8 months (Day 1 of Weeks 1, 5, 13, and 25, and 90 days after the last dose of monalizumab)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 15 | 9 | 36 | 33 | 31 | 18 | 17 | 18 | 30 | 2 | 39 | 1
Participants
  Persistent Positive | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Transient Positive | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-boosted ADA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-emergent ADA | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Positive ADA to Cetuximab
Description: Number of participants with positive ADA to cetuximab are reported. Persistent positive is defined as positive at >= 2 post-baseline assessments (with >=16 weeks between first and last positive) or positive at last post-baseline assessment. Transient positive is defined as negative at last post-baseline assessment and positive at only one post-baseline assessment or at >= 2 post-baseline assessments (with <16 weeks between first and last positive). Treatment-boosted ADA is defined as baseline ADA titer that was boosted to a 4-fold or higher level following drug administration. Treatment-emergent ADA is defined as the sum of treatment-induced ADA (post-baseline positive only) and treatment-boosted ADA.
Time Frame: Day 1 through 54.8 months (Day 1 of Weeks 1, 5, 9 [if EOT occurred], and 13, and 30 days after the last dose of monalizumab)
Population: as for outcome 25
Measure: Count of Participants; unit: Participants
Arm/Group | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 18 | 28 | 35 | 1 | 0
Participants
  Persistent Positive | 0 | 1 | 0 | 0 | 0
  Transient Positive | 0 | 0 | 0 | 0 | 0
  Treatment-boosted ADA | 0 | 0 | 0 | 0 | 0
  Treatment-emergent ADA | 0 | 1 | 0 | 0 | 0

28. Secondary Outcome: Number of Participants With Programmed Death Ligand 1 (PD-L1) Expression in Pretreatment Tumor Biopsies
Description: Number of participants with PD-L1 expression in pre-treatment tumor biopsies is reported. The participants were stratified into four categories: tumor cells (TC) >= 25%, TC<25%, TC>=1%, and TC<1%, based on the historical use of PD-L1 cutoffs.
Time Frame: Screening (Days -28 to -1)
Population: As-treated population included participant who received any study drugs and were analyzed according to the treatment they actually received. Here, number of participants analyzed (N) denotes those participants for whom PD-L1 testing was performed and number analyzed (n) denotes those participants for whom PD-L1 status was obtained.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 13 | 14 | 29 | 37 | 32 | 16 | 16 | 18 | 31 | 33 | 36 | 32
Participants
  TC>=25% | 0 | 0 | 0 | 2 | 1 | 0 | 5 | 1 | 6 | 0 | 0 | 0 | 1 | 1 | 0
  TC<25% | 3 | 3 | 3 | 11 | 13 | 29 | 32 | 31 | 10 | 16 | 18 | 31 | 32 | 35 | 32
  TC>=1% | 1 | 1 | 1 | 6 | 2 | 5 | 22 | 16 | 8 | 3 | 0 | 5 | 7 | 7 | 5
  TC<1% | 2 | 2 | 2 | 7 | 12 | 24 | 15 | 16 | 8 | 13 | 18 | 26 | 26 | 29 | 27

29. Secondary Outcome: Number of Participants With Human Leukocyte Antigen (HLA)-E Expression in Pretreatment Tumor Biopsies
Description: The HLA-E expression in pre-treatment tumor biopsies is reported.
Time Frame: Screening (Days -28 to -1)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
Number analyzed (Participants) | 3 | 3 | 3 | 18 | 18 | 40 | 40 | 40 | 20 | 18 | 18 | 39 | 41 | 44 | 37
Participants
  HLA-E Carcinoma | 3 | 3 | 3 | 12 | 13 | 28 | 36 | 32 | 16 | 16 | 17 | 30 | 33 | 34 | 32
  HLA-E Lymphocyte | 3 | 3 | 3 | 12 | 13 | 30 | 37 | 32 | 17 | 16 | 17 | 29 | 32 | 34 | 32
  HLA-E Endothelium | 3 | 3 | 3 | 13 | 13 | 30 | 37 | 33 | 17 | 16 | 17 | 30 | 31 | 34 | 32

ADVERSE EVENTS:
Time Frame: Day 1 through 246.9 weeks (maximum observed duration)
Description: All-cause mortality data was analyzed as per ITT population, and AE/SAE data was analyzed as per As-treated population.
Arm/Group | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/3 | 0/3 | 16/18 | 14/18 | 29/40 | 34/40 | 28/40 | 19/20 | 10/18 | 8/18 | 29/40 | 29/41 | 29/44 | 27/37
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 1/3 | 8/18 | 4/18 | 11/40 | 16/40 | 17/40 | 7/20 | 10/18 | 11/18 | 10/39 | 5/41 | 9/44 | 11/37
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 18/18 | 16/18 | 39/40 | 40/40 | 39/40 | 20/20 | 18/18 | 18/18 | 39/39 | 41/41 | 44/44 | 36/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W (N=3) | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W (N=3) | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W (N=3) | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (N=18) | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W (N=18) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) (N=40) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) (N=40) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) (N=40) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) (N=20) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W (N=18) | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W (N=18) | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W (N=39) | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W (N=41) | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W (N=44) | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W (N=37)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (3) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalation Cohort 1: Monalizumab 22.5 mg Q2W + Durvalumab 1500 mg Q4W (N=3) | Dose-escalation Cohort 2: Monalizumab 75 mg Q2W + Durvalumab 1500 mg Q4W (N=3) | Dose-escalation Cohort 3: Monalizumab 225 mg Q2W + Durvalumab 1500 mg Q4W (N=3) | Dose-escalation Cohort 4: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (N=18) | Dose-escalation Cohort 5: Monalizumab 750 mg Q4W + Durvalumab 1500 mg Q4W (N=18) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (MSS-CRC) (N=40) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Ovarian) (N=40) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (Endometrial MSS) (N=40) | Dose-expansion Cohort: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W (NSCLC) (N=20) | Exploration Cohort A1: Monalizumab 750 mg Q2W+Durvalumab 1500 mg Q4W+mFOLFOX6 Q2W+Bevacizumab Q2W (N=18) | Exploration CohortA2: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + mFOLFOX6 Q2W + Cetuximab Q2W (N=18) | Exploration Cohort C1A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W (N=39) | Exploration Cohort C1B: Monalizumab 750 mg Q2W + Cetuximab Q2W (N=41) | Exploration Cohort C2A: Monalizumab 750 mg Q2W + Durvalumab 1500 mg Q4W + Cetuximab Q2W (N=44) | Exploration Cohort C2B: Monalizumab 750 mg Q2W + Cetuximab Q2W (N=37)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 4 (7) | 4 (4) | 9 (10) | 13 (17) | 16 (17) | 3 (4) | 12 (26) | 10 (10) | 9 (12) | 8 (9) | 8 (9) | 7 (8)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal discharge (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal tenesmus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (7) | 3 (3) | 1 (1) | 6 (8) | 3 (3)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (9) | 1 (1) | 8 (13) | 10 (10) | 6 (7) | 4 (4) | 7 (8) | 3 (3) | 7 (9) | 8 (8) | 7 (8) | 1 (1)
Administration site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adverse drug reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 5 (5) | 2 (3) | 12 (13) | 2 (3) | 10 (21) | 1 (1) | 1 (1) | 2 (3) | 3 (4) | 0 (0) | 4 (4)
Catheter site dermatitis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site erosion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 1 (1) | 5 (5) | 3 (3) | 8 (11) | 2 (2)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (3) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 7 (7) | 11 (11) | 20 (22) | 1 (1) | 14 (33) | 7 (9) | 14 (20) | 8 (9) | 11 (15) | 6 (6)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 2 (4) | 1 (1)
Injection site discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (4) | 4 (4) | 4 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (1) | 5 (5) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 8 (9) | 8 (12) | 6 (6) | 2 (2) | 6 (9) | 4 (4) | 14 (17) | 6 (9) | 15 (18) | 6 (8)
Secretion discharge (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Xerosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (5) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conduction disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related hypersensitivity reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bacteriuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Clostridium bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 10 (10) | 9 (11) | 1 (1) | 3 (7) | 2 (4) | 6 (7) | 1 (1) | 4 (4) | 4 (5)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Oral fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 4 (4) | 4 (4) | 6 (6)
Penile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 7 (9) | 3 (3) | 0 (0) | 4 (6) | 1 (1) | 3 (3) | 4 (4) | 3 (3) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (3) | 9 (9) | 9 (12) | 4 (4)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (3) | 3 (4) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 5 (5) | 4 (4)
Amylase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (7) | 7 (14) | 3 (3) | 1 (3) | 5 (6) | 4 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 3 (3) | 4 (4) | 3 (4) | 2 (2) | 0 (0) | 5 (6) | 4 (4) | 6 (6) | 8 (11) | 8 (8) | 6 (10)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 3 (3) | 4 (4) | 5 (7) | 4 (4)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (3) | 4 (7) | 4 (4) | 2 (5) | 4 (5)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (4)
Blood creatine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 7 (9) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 3 (4)
Blood fibrinogen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood uric acid decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carbohydrate antigen 125 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 3 (3) | 3 (4) | 2 (2) | 5 (5) | 3 (3) | 5 (7)
General physical condition abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 2 (2)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 9 (14) | 2 (2) | 3 (5) | 8 (9) | 6 (14)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 1 (1) | 3 (3) | 3 (3) | 5 (10)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 5 (7) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tri-iodothyronine free decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin i increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 4 (6) | 3 (3)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
White blood cells urine positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adult failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 4 (4) | 7 (9) | 5 (5) | 14 (14) | 3 (3) | 8 (11) | 5 (6) | 10 (11) | 5 (6) | 9 (9) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercreatininaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (4) | 1 (1)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 2 (2) | 1 (2) | 3 (3) | 1 (2) | 3 (6)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 4 (4) | 3 (4) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (8) | 3 (4)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 4 (6) | 0 (0) | 3 (3) | 2 (3) | 2 (2) | 2 (2) | 5 (7) | 5 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 5 (7) | 3 (3) | 0 (0) | 1 (1) | 4 (7) | 3 (4) | 8 (8) | 9 (13) | 10 (21)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 3 (4) | 0 (0) | 2 (3) | 1 (3) | 2 (3) | 6 (8) | 5 (5) | 4 (5)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polydipsia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 4 (5) | 6 (7) | 4 (4) | 5 (5) | 3 (3) | 2 (5) | 3 (4) | 2 (3) | 4 (4) | 4 (4) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (16) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 6 (6) | 5 (5) | 6 (6) | 1 (1) | 3 (4) | 2 (2) | 4 (4) | 5 (5) | 6 (7) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Euthyroid sick syndrome (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 4 (4) | 1 (1) | 2 (3) | 2 (3) | 0 (0) | 6 (6) | 0 (0) | 9 (10) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 6 (7) | 5 (7)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Central nervous system necrosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 5 (5) | 1 (1) | 6 (7) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 2 (2)
Dysaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thyroid mass (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalomalacia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 7 (8) | 0 (0) | 4 (5) | 1 (1) | 6 (7) | 0 (0) | 8 (9) | 17 (19) | 12 (13) | 8 (9)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lhermitte's sign (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 10 (12) | 11 (14) | 1 (1) | 1 (1) | 1 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amaurosis fugax (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hallucinations, mixed (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 1 (1) | 4 (4) | 0 (0) | 2 (6) | 1 (1) | 3 (3) | 3 (3) | 5 (5) | 4 (4)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mood swings (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nightmare (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blepharospasm (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder irritation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chromaturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (5)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Scrotal dermatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (5) | 5 (6) | 6 (7) | 6 (6) | 9 (10) | 2 (3) | 3 (3) | 5 (7) | 4 (4) | 2 (2) | 4 (5)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 6 (6) | 6 (6) | 6 (7) | 6 (6) | 5 (12) | 1 (2) | 5 (6) | 4 (4) | 5 (5) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 5 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 8 (15) | 20 (21) | 24 (24) | 28 (41) | 23 (25)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelids pruritus (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 5 (5) | 2 (2) | 5 (5) | 3 (3) | 10 (10)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intertrigo (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Onychalgia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (3) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 3 (3) | 7 (7) | 1 (1) | 3 (3) | 4 (8) | 6 (6) | 8 (10) | 12 (15) | 7 (11)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 4 (4) | 5 (5) | 3 (4) | 3 (3) | 1 (1) | 3 (3) | 9 (14) | 12 (14) | 8 (8) | 5 (9) | 9 (9)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (8) | 6 (6) | 5 (5) | 4 (6) | 4 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trichorrhexis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central venous catheterisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 6 (7) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (3) | 2 (2) | 3 (3) | 10 (10) | 8 (9) | 5 (5) | 0 (0) | 4 (4) | 6 (6) | 5 (5) | 7 (7) | 7 (7) | 2 (2)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Abdominal rigidity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 8 (15) | 6 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 9 (9) | 2 (2) | 7 (8) | 9 (9) | 4 (4) | 2 (2) | 5 (5) | 3 (3) | 4 (5) | 7 (8) | 10 (12) | 1 (1)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (1) | 5 (5) | 2 (2) | 6 (6) | 10 (12) | 10 (11) | 6 (7) | 8 (24) | 6 (8) | 5 (8) | 5 (7) | 9 (12) | 7 (10)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2021-05-31): https://cdn.clinicaltrials.gov/large-docs/35/NCT02671435/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/35/NCT02671435/SAP_005.pdf